CLINICAL TRIAL: NCT03701750
Title: Effect of Low-Molecular-Weight-Heparin (LMWH) on Pregnancy Outcome in Women With Multiple Failures of IVF-ET
Brief Title: Effect of LMWH on Pregnancy Outcome in Women With Multiple Failures of IVF-ET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Zhongshan Urology Hospital (Other Government)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yong Zeng, Head of Hospital, Shenzhen Zhongshan Urology Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: szuh-2018-CT001
Record Dates: First submitted 2018-10-07; First posted 2018-10-10 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Infertility
Keywords: IVF; pregnancy; LMWH; Low Molecular Weight Heparin; Assisted Reproductive Technology; Implantation
MeSH Terms: conditions — Infertility | interventions — Heparin, Low-Molecular-Weight; enoxaparin sodium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Low Molecular Weight Heparin (enoxaparin sodium) + routine luteal phase support
  Interventions: Drug: Low Molecular Weight Heparin (enoxaparin sodium)
- Control Arm (No Intervention): routine luteal phase support

INTERVENTIONS:
Drug: Low Molecular Weight Heparin (enoxaparin sodium) — enoxaparin sodium 40mg/day subcutaneously after oocyte collection, and routine luteal phase support after embryo transfer until clinical pregnancy confirmed by ultrasound
  Arms: Experimental Arm

SUMMARY:
Low-Molecular-Weight-Heparin (LMWH) has been used empirically in patients undergoing in-vitro fertilization embryo transfer (IVF-ET) with the purpose to aid in improving pregnancy outcomes. The potential mechanism is that LMWH could exert its anticoagulant effect by inhibiting factor Xa, reducing the risk of insufficiency blood supply in the very early stage of pregnancy. Moreover, LMWH is supposed to play a role in manipulating blastocyst supposition, adhesion, and implantation, as well as trophoblast differentiation and invasion. However, limited high-quality clinical trials focus on the effectivity of LMWH in IVF-ET, and the published evidence is not consensus, leading to considerable controversy in the clinical application of LMWH in IVF-ET patients. Here, investigators try to evaluate the effect of LMWH on pregnancy outcome in women with multiple failures of IVF-ET via a multi-center randomized controlled trial.

DETAILED DESCRIPTION:
Implantation failure seems to be inevitable in some couples undergoing IVF-ET treatment, despite transferred with high-quality embryos. There are several factors, including coagulation, are supposed to contribute to the implantation failure. Several groups reported that inherited and acquired coagulation is highly prevalent in women with recurrent implantation failure (RIF). Besides, women undergoing assisted reproduction are more likely to expose to thrombotic risks because high-dose exogenous gonadotrophins are given to harvest more oocytes for the fertilization. Given the risk of thrombosis, patients are often recommended to receive thromboprophylaxis with unfractionated heparin (UFH) or low molecular weight heparin (LMWH) in many clinics empirically.

LMWH is generated by depolymerization from UFH. Compared with UFH, LWMH exerts its anticoagulant effect mainly by inhibiting factor Xa rather than factor IIa. LMWH has a more predictable antithrombotic response and allows the administration to patients themselves without the laboratory monitoring. Also, it substantially reduces the risk of heparin-induced thrombocytopenia (HIT).

Beyond its anticoagulant effects, heparin is supposed to improve pregnancy outcomes by modulating blastocyst supposition, adhesion and implantation and as well as trophoblast differentiation and invasion through interactions with several adhesion molecules, growth factors, cytokines, and enzymes. Also, complement activation induced by aPL antibodies in mice is inhibited, and pregnancy complications are attenuated when treated with heparin.

Unfortunately, the use of LMWH in IVF/ET seems based on biological plausibility rather than evidence of efficacy. The high-quality studies (randomized controlled trials or prospective controlled trials) are limited, and the results are controversial. A meta-analysis (including 2 RCT and 1 quasi-RCT) reported that there is no difference in implantation rate in women with ≥3 recurrent implantation failure when treated with LMWH. Although live birth rate (LBR) and miscarriage rates are improved, investigators are still concerned because limited studies and patients were included in this analysis. Even in the non-RIF patients with or without thrombophilia defects, no consensus results could be achieved.

Given the burden of daily injection, skin irritation at injection site and other potential side-effects, the effectivity of LMWH in IVF/ET should be carefully examined even though LMWH is regarded as safe thromboprophylaxis. Hence, investigators propose a multi-center randomized study to evaluate the efficacy of Heparin in IVF-ET.

ELIGIBILITY:
Inclusion Criteria:

* ≥2 consecutive IVF/ICSI-ET without clinical pregnancy
* ≥2 oocytes retrieval cycles
* 19<BMI≤25
* Normal ovarian reserve ( AMH> 1, FSH <10 )
* Willing and able to sign the informed consent.

Exclusion Criteria:

* Uterine abnormalities confirmed by hysterosalpingography or hysteroscopy
* Parental chromosomal abnormalities
* PCOS
* Anti-phospholipid Syndrome
* Endocrine disorder
* Endometriosis
* Hydrosalpinx
* Chronic disease (liver, renal, thyroid, and thrombocytopenia)
* Regular anticoagulation or antiplatelet treatment
* Patients who had contraindication for unfractionated heparin therapy
* History of tuberculosis, HIV, HBV, HCV or tests indicating carriage of HBV or HCV, or positive interferon-gamma release assay in any of the couple
* Enrollment in another clinical trial

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Time of delivery up to 42 weeks gestation
  Birth of liveborn

SECONDARY OUTCOMES:
Embryo implantation rate | 4 weeks
  Gestational sacs are seen by ultrasound
Clinical pregnancy rate | 7-8 weeks
  Fetal heartbeat is seen by ultrasound
Miscarriage rate | Up to 28 weeks
  After clinical pregnancy confirmed, before 28 weeks
Ovarian hyperstimulation syndrome (OHSS) rate | Up to 3 weeks after COH
  Ovarian hyperstimulations syndrome after COH

CONTACTS AND LOCATIONS:
Overall Officials: Haixiang Sun, M.D. Ph.D, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Jing Yang, M.D. Ph.D, Principal Investigator — Renmin Hospital of Wuhan University; Ruochun Lian, M.D. Ph.D, Principal Investigator — Shenzhen Zhongshan Urology Hospital
Locations (3):
- China (3):
  - Clinical Research Center for Reproductive Medicine, Fertility Center, Shenzhen Zhongshan Urology Hospital, Shenzhen, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Urman B, Ata B, Yakin K, Alatas C, Aksoy S, Mercan R, Balaban B. Luteal phase empirical low molecular weight heparin administration in patients with failed ICSI embryo transfer cycles: a randomized open-labeled pilot trial. Hum Reprod. 2009 Jul;24(7):1640-7. doi: 10.1093/humrep/dep086. Epub 2009 Apr 8. PMID 19357135
- [Background] Noci I, Milanini MN, Ruggiero M, Papini F, Fuzzi B, Artini PG. Effect of dalteparin sodium administration on IVF outcome in non-thrombophilic young women: a pilot study. Reprod Biomed Online. 2011 Jun;22(6):615-20. doi: 10.1016/j.rbmo.2011.03.016. Epub 2011 Mar 22. PMID 21498125
- [Background] Stern C, Chamley L, Norris H, Hale L, Baker HW. A randomized, double-blind, placebo-controlled trial of heparin and aspirin for women with in vitro fertilization implantation failure and antiphospholipid or antinuclear antibodies. Fertil Steril. 2003 Aug;80(2):376-83. doi: 10.1016/s0015-0282(03)00610-1. PMID 12909502